CLINICAL TRIAL: NCT01207999
Title: Human Papillomavirus (HPV) Type Distribution in Adult African Women Diagnosed With Invasive Cervical Cancer
Brief Title: Type Distribution of Human Papillomavirus in Adult African Women Diagnosed With Invasive Cervical Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Cape Town (Other); African Organization for Research and Training in Cancer (AORTIC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 109117
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Infections, Papillomavirus; Cervical Cancer
Keywords: Human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cervical specimen

GROUPS / COHORTS (1):
- Group A: Subjects diagnosed with invasive cervical cancer
  Interventions: Procedure: Collection of cervical cancer tissue samples; Other: Data collection

INTERVENTIONS:
Procedure: Collection of cervical cancer tissue samples — Cervical samples will be tested for histopathology diagnosis and human papillomavirus DNA testing.
Other: Data collection — Questionnaire completion

SUMMARY:
The aim of the study is to assess the distribution of the most frequent types of human papillomavirus in African women diagnosed with invasive cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* A female aged 21 years or more, presenting with a lesion macroscopically suggestive of invasive cervical cancer.
* Scheduled for cervical biopsy as per routine procedure at the participating institution on the day of the visit or on a later date.
* Written or oral-witnessed informed consent obtained from the subject prior to any study procedure.
* No prior chemo- or radiotherapy for cervical cancer.

Exclusion Criteria:

Not applicable

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged ≥ 21 years at the time the cervical specimen is taken, diagnosed with cervical lesion macroscopically suggestive of invasive cervical cancer, scheduled for cervical biopsy as per routine procedure.
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of any of the human papillomavirus types (HPV-16, 18, 31, 33, 35, 45, 52 and 58) among the women diagnosed with invasive cervical cancer | Average time frame: 6-12 months
Occurrence of any of the human papillomavirus types (human papillomavirus-16, 18, 31, 33, 35, 45, 52 and 58) among the women diagnosed with squamous cell carcinoma | Average time frame: 6-12 months

SECONDARY OUTCOMES:
Proportion of squamous cell carcinoma cases versus adenocarcinoma and other histologic tumour types of invasive cancer among the women diagnosed with invasive cervical cancer | Average time frame:6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Ghana (2):
  - GSK Investigational Site, Accra
  - GSK Investigational Site, Kumasi
- Nigeria (2):
  - GSK Investigational Site, Ibadan
  - GSK Investigational Site, Lagos
- GSK Investigational Site, Observatory, Western Province, South Africa